CLINICAL TRIAL: NCT06423040
Title: Exploring the Effectiveness of Applying Social Media Chatbot for Providing Real-Time Feedback on Physical Activity Education for Older Adults
Brief Title: Social Media Chatbot on Physical Activity Education for Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202403043
Record Dates: First submitted 2024-05-08; First posted 2024-05-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-04

CONDITIONS: Exercise; Self Efficacy; Behavioral Regulation; Healthy Aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Experiment (Experimental)
  Interventions: Other: Social Media Chatbot on Physical Activity Education

INTERVENTIONS:
Other: Social Media Chatbot on Physical Activity Education — a social media chatbot was used to provide a continuous and real-time multimedia health education program on physical activity for the older adults, as well as supportive messages and feedbacks.
  Arms: Experiment

SUMMARY:
In this study, a social media chatbot was used to provide a continuous and real-time multimedia health education program on physical activity for the older adults, as well as supportive messages and feedbacks, to improve physical activity and exercise self-efficacy among the older adults. This study was a cluster randomized trial, and participants were recruited from community care stations and activity centers in Taipei City. The experimental group was involved in an 8-week, 5-day-a-week intervention with a total of 40 multimedia physical activity education programs, and users were provided with real-time feedback interactions and regular physical activity education guidelines, and self-administered questionnaires were used for data collection. The research instruments include basic personal information, International Physical Activity Questionnaire, Exercise Self-Efficacy Scale, Behavioral regulation in exercise questionnaire-2, Exercise Benefits/Barriers Scale, and the statistical methods will be descriptive statistics, independent sample t-test, paired sample t-test, and one-way analysis of covariance.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 60 to 85 years old living in Taipei City, healthy or with chronic conditions
2. Those who can listen, read and write Chinese
3. Those who have used smartphones in the past month and can use Line social software
4. Those who voluntarily participate in this study, can understand the research content after explanation and explanation, and sign the subject consent form

Exclusion Criteria:

1. Those who are advised by a doctor not to exercise
2. Those who must exercise under the supervision of medical personnel
3. Patients with severe cardiovascular disease
4. Anyone with disability or cognitive impairment
5. Persons living in long-term care institutions

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Physical activity | up to 8 weeks
  International Physical Activity Questionnaire
Self-Efficacy | up to 8 weeks
  Exercise Self-Efficacy Scale
Behavioral regulation | up to 8 weeks
  Behavioral regulation in exercise questionnaire-2
Benefits/Barriers | up to 8 weeks
  Exercise Benefits/Barriers Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No